CLINICAL TRIAL: NCT01527409
Title: The Efficacy of Health Partnership Program for Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); Korea University Anam Hospital (Other); Asan Medical Center (Other); Ajou University School of Medicine (Other); Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, YoungSung Lee, Head, Division of Cancer Management Branch, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCCCTS-11-598
Record Dates: First submitted 2012-01-10; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer; Colon Cancer; Gastric Cancer; Lung Cancer
Keywords: Exercise; Diet; Posttraumatic growth
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Lung Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimetal Arm (Experimental): Providing tailored health care program, which provides various information related to exercise, diet, and posttraumatic growth.
  Tailored health partnership program consists of three strategic areas (exercise, diet, and posttraumatic growth). Those areas are based on the transtheoretical model (TTM), social cognitive theory, PRECEDE-PROCEED model, and Health behavior model.
  Patients who participate in the tailored health partnership program will be received tailored manual and workbook for tele-coaching that help them to lead their healthy life.
  Also, patients will be provided a workshop for leadership that is dealt with controlling their healthy life.
  Interventions: Behavioral: Tailored health partnership program
- Control Arm (No Intervention): Providing usual care. Also, patients will be provided a workshop for health education that is dealt with ten areas (smoke and drinking, diet, exercise, posttraumatic growth, distress, pain, comorbidity, sleep disturbance, pain, and energy conservation).
  Twelve month later, patients will be provided the tailored health partnership program which is especially dealing with exercise, diet, and posttraumatic growth.
  Interventions: Behavioral: Usual care and health education workshop

INTERVENTIONS:
Behavioral: Tailored health partnership program — When intervention group participate in the tailored program, they can receive various information which is related with three strategic areas (exercise, diet, and posttraumatic growth).
  Three areas are based on the transtheoretical model (TTM), social cognitive theory, PRECEDE-PROCEED model, and Health behavior model.
  Patients will be received tailored manual and workbook for health tele-coaching that help them to lead their healthy life.
  The health tele-coaching will be operated sixteen times for 24 weeks. Intervention group will be provided three contents (exercise, diet, and posttraumatic growth) from health partners. The health partners took a certificate that is related with health, leadership and coaching.
  Also, patients will be provided a workshop for leadership that is dealt with controlling their healthy life. It will be proceeded for four hours. Three hours is for the leadership, and the last one hour is for presentation of their health mission statement.
  Arms: Experimetal Arm
Behavioral: Usual care and health education workshop — While intervention group participate in the tailored health partnership program, control group can receive various information which is related with ten contents for health management (smoke and drinking, diet, exercise, posttraumatic growth, distress, pain, comorbidity, sleep disturbance, pain, and energy conservation). They will be provided a workshop and booklet for a health education for four hours.
  Twelve month later, they will be provided the tailored health partnership program which is especially dealing with exercise, diet, and posttraumatic growth as same as the intervention group.
  Arms: Control Arm

SUMMARY:
The Objectives of this study is

1. To evaluate the efficacy for exercise, diet, and posttraumatic growth as a result of participating in tailored program (Health Partnership Program) for 24 weeks
2. To evaluate the efficacy for quality of life, life satisfaction, health leadership, anxiety, depression, impact of event, social support, cancer belief as a result of participating in tailored program (Health Partnership Program) for 24 weeks
3. To assess the efficacy of such intervention compared with usual care in cancer patients

DETAILED DESCRIPTION:
***Background

Improving cancer patients' quality of life has been increasing subject of research for several years. Especially, the patients and their families who are needed to deal with specific care on diverse aspects, such as social, spiritual, existential, psychological aspect should be provided integrated program.

Multidimensional characteristics of the health partnership program were addressed in National Cancer Center (NCC) for exercise, diet, and posttraumatic growth based on transtheoretical (TTM) model, social cognitive theory, health behavioral model, and coaching strategies. This program points out the importance of behavioral approaches in managing their healthy life according to improve patterns of three areas (exercise, diet, and posttraumatic growth).

Strategies that investigators mentioned above can lead those three areas to be effective.

To objective of this study is to support cancer patients to cope with exercise, diet, and posttraumatic growth through tailored program (the health partnership program), and then evaluate the efficacy of the health partnership program.

From evidence extracted from a literature review, contents of the program was elaborated, and tailored from the TTM model. The curriculum is currently being reviewed and validated by expert group of oncologists, nurse, psychologist and health education scientists.

***Method

To determine the efficacy of the program (the health partnership program), a randomized controlled trial will be conducted:

After excluding patients with other causes (anemia, thyroid disease, co morbidities etc), 248 patients will be recruited based on statistical assumption of alpha (0.05), beta (0.20=power 80%), and dropout rate (15%).

First, patients will be stratified according to their age, sex (male vs. female), cancer types (stomach cancer, Breast cancer, cervical cancer, colorectal (except rectal cancer) cancer, and lung cancer), and then allocated to an intervention or control group.

When intervention group participates in the tailored program (the health partnership program), they can receive various information which is related to health management and improving quality of life.

The health partnership program consists of 16 time's tele-coaching, a self leadership workshop, and providing health materials (manuals, workbook, and booklet). Especially, those will be dealt with managing three areas; exercise, diet, and posttraumatic growth based on the transtheoretical model (TTM), social cognitive theory, health behavioral model, and coaching strategies.

Cancer patients who are participated in the tailored program will be received tailored feedbacks that enhance participants of the next level of the program.

On the other hand, the control group could not participate in the health partnership program. The control group could only be treated by usual care and a health education workshop with a health booklet. However, the control group can participate in the health partnership program after 12 month.

Data will be collected before randomization, after intervention, and after a follow-up of 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult(≥ 20 years)
* Within 24 months of completion of primary treatment with curative intent (Surgery, radiotherapy, chemotherapy)
* Breast, cervical, colorectal (except rectal cancer), lung, and stomach cancer
* More than two problematic areas among exercise, diet (Fruit & Vegetable: F&V), and posttraumatic growth(exercise < 150min/week, ≥ 3mets, F&V < 5/day, PTGI < 71)

Exclusion Criteria:

* Evidence of secondary tumor, metastasis and recurrence
* Patients undergoing or planning surgery, radiation therapy or chemotherapy
* Not Korean speaking and reading (Not communication with Korean)
* Not understanding of the study purpose and not written informed consent
* Participants who have an similar study experience
* Major health problem in which exercise/nutrition intervention is contraindicated at the discretion of clinician; cardiovascular disease (congestive heart failure, angina), pulmonary disease (chronic obstructive pulmonary disease, restrictive pulmonary disease), uncontrolled hypertension, poorly controlled diabetes and severe musculoskeletal disease and so on
* Sign of infection (body temperature ≥ 37.2℃ or WBC ≥ 11,000)
* Being pregnant
* Thrombocytopenia (platelet count ≤ 100,000/mcl)
* Anemia (Hb ≤ 10g/dL)
* SGOT or SGPT > 40 IU/L
* Creatinine > 1.2 mg/dL
* Severe psychiatric disorder (psychotic disorder, major depression and so on) or suicidal tendencies
* dyspnea

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Exercise, Diet, and Posttraumatic Growth Inventory(PTGI) | baseline, 3month, 6month, and 12month
  How much the patient does exercise will be measured using "MET" score. Change in diet will be observed by analyzing 3day recall.

SECONDARY OUTCOMES:
Seven habit profile | baseline, 3month, 6month, and 12month
the European Organisation for the Research and Treatment of Cancer Quality-of-life Questionnaire-Core 30(EORTC QLQ C-30) | baseline, after 3month, 6month, and 12month
Ed Diner's Satisfaction with Life Scale | baseline, after 3month, 6month, and 12month
Impact of Event Scale-Revised | baseline, after 3month, 6month, and 12month
Social Support(MOS-SSS) | baseline, after 3month, 6month, and 12month
the Hospital Anxiety and Depression scale(HADS) | baseline, after 3month, 6month, and 12month
Cancer Belief System(CBS) | baseline, after 3month, 6month, and 12month

CONTACTS AND LOCATIONS:
Overall Officials: YoungSung Lee, MD, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (10):
- South Korea (10):
  - Seoul National University Boondang Hospital, Boondang, Gyunggi
  - National Cancer Center, Goyang, Gyunggi
  - Ajou University Medical Center, Suwon, Gyunggi
  - Keimyng University Dongsan Center, Daegu
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Eun Sook Lee, M. K. L., Soo Hyun Kim, Jung Sil Ro, Han Sung Kang, Seok Won Kim, Keun Seok Lee, Young Ho Yun. (2010(Accepted) ).
- [Background] Kravitz, R. L., D. J. Tancredi, et al. (2009).
- [Background] Park, S. M., M. K. Lim, et al. (2007).
- [Background] Shin, H. W., D. Y. Noh, et al. (2009).
- [Background] Soo Hyun Kim, M. S. S., Han Sul Lee, Eun Sook Lee, Jung Sil Ro, Han Sung Kang, Seok Won Kim, Won Hee Lee, Chun Ja Kim, Hee Soon Kim, Joo hyung Kim, Young Ho Yun (2010).
- [Background] Street, R. L., Jr., C. Slee, et al.
- [Background] Vale, M. J., M. V. Jelinek, et al. (2003).
- [Background] Wolever, R. Q., M. Dreusicke, et al.
- [Background] Demark-Wahnefried W, Clipp EC, Lipkus IM, Lobach D, Snyder DC, Sloane R, Peterson B, Macri JM, Rock CL, McBride CM, Kraus WE. Main outcomes of the FRESH START trial: a sequentially tailored, diet and exercise mailed print intervention among breast and prostate cancer survivors. J Clin Oncol. 2007 Jul 1;25(19):2709-18. doi: 10.1200/JCO.2007.10.7094. PMID 17602076
- [Background] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455
- [Background] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Background] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Background] Kim SH, Shin MS, Lee HS, Lee ES, Ro JS, Kang HS, Kim SW, Lee WH, Kim HS, Kim CJ, Kim J, Yun YH. Randomized pilot test of a simultaneous stage-matched exercise and diet intervention for breast cancer survivors. Oncol Nurs Forum. 2011 Mar;38(2):E97-106. doi: 10.1188/11.ONF.E97-E106. PMID 21356647
- [Derived] Yun YH, Kim YA, Lee MK, Sim JA, Nam BH, Kim S, Lee ES, Noh DY, Lim JY, Kim S, Kim SY, Cho CH, Jung KH, Chun M, Lee SN, Park KH, Park S. A randomized controlled trial of physical activity, dietary habit, and distress management with the Leadership and Coaching for Health (LEACH) program for disease-free cancer survivors. BMC Cancer. 2017 May 2;17(1):298. doi: 10.1186/s12885-017-3290-9. PMID 28464804